CLINICAL TRIAL: NCT03984240
Title: The Effects of Mild Sedation on Compensatory Upper Limb Motor Function Networks Based on Multimodal Magnetic Resonance Imaging in With Gliomas in Brain Eloquent Areas
Brief Title: The Effects of Mild Sedation on Motor Function Networks in Patients With Brian Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Nan Lin, Principal Investigator, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81701038
Record Dates: First submitted 2019-06-08; First posted 2019-06-12 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2023-07

CONDITIONS: Brain Glioma; Midazolam; Dexmedetomidine
Keywords: functional MRI; Sensory Motor Function; Midazolam; Mild sedation; Dexmedetomidine
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frontal-Parietal Supratentorial Brain Glioma Group (Experimental): The frontal-parietal brain area glioma being diagnosed by MRI scan.
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine
- control group (Active Comparator): Healthy volunteers without intracranial diseases.
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — Participant will be sedated by midazolam.
Drug: Dexmedetomidine — Participant will be sedated by dexmedetomidine.

SUMMARY:
It has been shown through functional MRI (Magnetic Resonance Imaging) that patients with gliomas in eloquent areas have compensated neurological function by virtue of brain post-injury reorganization. Our previous clinical research found that mild sedation could induce and/or exacerbate neurological deficits, especially in limb motor and ataxia function, in these patients presumably by impairing functional compensation,. Nevertheless it is still very unclear how mild sedation affects sensorimotor networks in brains where reorganization may be present. Since eloquent area glioma patients are frequently subjected to sedation, anesthetics, and neurological examinations perioperatively, it is important to investigate how mild sedation interacts with motor network reorganization and functional compensation. Our research in patients with eloquent area gliomas will utilize neurological evaluations and multimodal MRI to explore the changes in brain upper limb' motor network reorganization after mild sedation by different sedatives-anesthetics. The neurological evaluations include sensorimotor function scale and testing tool. Multimodal MRI consists of 3-dimentional structure, blood oxygen-level dependent for cortical activation and diffusion tensor imaging for subcortical conduction. The data from the clinical testing and functional MRI will be processed and analyzed along with other relevant clinical information. This research will answer the question of how mild sedation affects upper limb motor function networks in brains with eloquent area gliomas. This new information will help optimize perioperative anesthetic and sedative choice for patients with eloquent area gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 to 60 years old;
* Diagnosed as intracranial eloquent glioma by MRI, or healthy volunteer without any intracranial disease;
* Without history of chronic diseases;
* Without internal and/external metal object;
* Right handedness

Exclusion Criteria:

* Unable to cooperate the neurologic function evaluation;
* Neuropsychiatric disorders and/or taking antipsychotic medications;
* Drug and/or alcohol abuse;
* Receiving longterm sedatives and/or analgesics;
* Pregnant and/or lactation period patients;
* Present severe cardiovascular diseases;
* Having claustrophobia;
* Body mass index equal or more than 35 kg/m2;
* Anticipated difficult airway;
* History of severe obstructive sleep apnea;
* History of reflux

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Brain network connectivity | 2 hours following sedation
  will use fMRI and DTI

SECONDARY OUTCOMES:
upper limb's motor function | 2 hours following sedation
  will use 9-hole peg test and motor/sensory function evaluation
pathological diagnose of glioma | 2 weeks after surgery completion
  the detailed type of glioma and WHO glioma grade

CONTACTS AND LOCATIONS:
Overall Officials: Nan LIN, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No